CLINICAL TRIAL: NCT01510340
Title: Evaluation of a Tailored Virtual Intervention to Empower Persons Living With HIV for Therapy Self-management
Acronym: HIVMediconline
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CE 11.184
Record Dates: First submitted 2011-12-13; First posted 2012-01-16 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: HIV
Keywords: adherence; HIV; antiretroviral therapy; tailored web intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Web sites (No Intervention): Patients assigned to this arm are given a list of Web sites where they can collect information related to their condition at their leisure.
- VIH-TAVIE (Experimental): Patients assigned to this arm must follow the four interactive computer sessions
  Interventions: Behavioral: VIH-TAVIE

INTERVENTIONS:
Behavioral: VIH-TAVIE — The tailored virtual intervention is composed of four interactive computer sessions hosted by a virtual nurse who engages the PLHIV in a medication-intake self-management skills-learning process.
  Arms: VIH-TAVIE

SUMMARY:
The purpose of this study is to evaluate the efficacy of an online virtual intervention in optimizing adherence to antiretroviral medication intake among Persons Living with HIV (PLHIV).

ELIGIBILITY:
Inclusion Criteria:

* have to be under ART for at least six months¸
* have internet access

Exclusion Criteria:

* be pregnant
* active IV drug user
* actual diagnosis of psychiatric health problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2012-01; Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Adherence | 6 months
  Adherence will be evaluated through a self-administered questionnaire that was developed for and validated on the targeted population (Godin, Gagné, & Naccache, 2003). The questionnaire comprises seven items that serve to determine how many times a person forgets to take his or her medication. The questionnaire's validity was demonstrated (sensitivity: 71 %; specificity: 72%; correct classification: 72%; odds ratio: 6.15) using immunologic (CD4 count) and virologic (viral load) parameters as validation criteria. Adherence is defined as the intake of at least 95% of prescribed tablets.

CONTACTS AND LOCATIONS:
Overall Officials: José Côté, Ph.D., Principal Investigator — CRCHUM, Université de Montréal; Gaston Godin, Ph.D., Study Chair — Laval University; Yann-Gael Guéhéneuc, Ph.D., Study Chair — Polytechnique; Cécile Tremblay, MD,Ph.D., Study Chair — CRCHUM; Joanne Otis, Ph.D., Study Chair — Université du Québec a Montréal
Locations (1):
- José Côté, Montreal, Quebec, Canada

REFERENCES:
- [Result] Cote J, Rouleau G, Ramirez-Garcia MP, Auger P, Thomas R, Leblanc J. Effectiveness of a Web-Based Intervention to Support Medication Adherence Among People Living With HIV: Web-Based Randomized Controlled Trial. JMIR Public Health Surveill. 2020 Apr 20;6(2):e17733. doi: 10.2196/17733. PMID 32310145
- [Derived] Cote J, Godin G, Gueheneuc YG, Rouleau G, Ramirez-Garcia P, Otis J, Tremblay C, Fadel G. Evaluation of a real-time virtual intervention to empower persons living with HIV to use therapy self-management: study protocol for an online randomized controlled trial. Trials. 2012 Oct 5;13:187. doi: 10.1186/1745-6215-13-187. PMID 23039306
- See also: Related Info — http://www.crsi.umontreal.ca